CLINICAL TRIAL: NCT06567912
Title: The Development of the Simulation Curriculum and Artificial Intelligence-incorporated Assessment Tools for Transesophageal Echocardiography in Patients With Cardiac Arrest
Brief Title: The Development of the Simulation Curriculum and AI-incorporated Assessment Tool for Transesophageal Echocardiography
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202211107RINB
Record Dates: First submitted 2024-08-18; First posted 2024-08-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: TEE simulation curriculum — The curriculum comprised of one-hour lecture and 3-hour hands-on training on a simulation model.

SUMMARY:
This study aims to establish a novel transesophageal echocardiography (TEE) simulation curriculum based on previous research results and suggestions from the American College of Emergency Physicians. To better evaluate the efficacy of the curriculum, an evaluation model utilizing artificial intelligence (AI) would be introduced. The study population is at least 60 junior physicians in the emergency department or other departments interested in TEE. After the curriculum, junior physicians could utilize TEE on cardiac arrest patients and improve diagnostic accuracy and patient outcomes.

DETAILED DESCRIPTION:
This study aims to establish a novel TEE simulation curriculum based on previous research results and suggestions from the American College of Emergency Physicians. To better evaluate the efficacy of the curriculum, an evaluation model utilizing artificial intelligence (AI) would be introduced. The study population is at least 60 junior physicians in the emergency department or other departments interested in TEE. After the curriculum, junior physicians could utilize TEE on cardiac arrest patients and improve diagnostic accuracy and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Emergency physicians interested in TEE learning.

Exclusion Criteria:

Emergency physicians are not interested in TEE learning.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: emergency physicians
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
learning outcomes:immediate assessment | 4 hours
  image acquisition and image quality using 5-point Likert scales. The range from 1 (the worst) to 5 (the best).
learning outcomes: 3-month evaluation | 3 months
  image acquisition and image quality using 5-point Likert scales. The range from 1 (the worst) to 5 (the best).
the efficiency of AI model | 6 months
  the AI model to recognize the TEE views, including sensitivity, specificity, PPV, NPV

CONTACTS AND LOCATIONS:
Locations (1):
- Lien, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No